CLINICAL TRIAL: NCT03768336
Title: A Stress Management and Resiliency Program for Adolescent and Young Adult Cancer Survivors
Brief Title: A Stress Management and Resiliency Program for Adolescent and Young Adult Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Giselle K. Perez Lougee, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-428; 1K07CA211955-01A1 (NIH)
Record Dates: First submitted 2018-12-04; First posted 2018-12-07 (Actual); Results first posted 2022-12-28 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: Cancer; Behavioral Intervention; Adolescent; Young Adult
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist Control (Active Comparator): * The 3RP-AYA will be delivered in weekly sessions over the course of approximately 8 weeks, for a total of 8 sessions
  * Mini relaxation practice
  * Weekly goal check-ins
  * RR-practice
  Interventions: Other: Waitlist control
- 3RP Group Sessions (Experimental): * The 3RP-AYA will be delivered in weekly sessions over the course of approximately 8 weeks, for a total of 8 sessions
  * Mini relaxation practice
  * Weekly goal check-ins
  * RR-practice
  Interventions: Other: 3RP-AYA

INTERVENTIONS:
Other: Waitlist control — The 3RP is a group program that-through a variety of mind-body approaches, such as imagery, relaxation, and yoga-seeks to buffer stress and promote psychological resiliency and physical well-being. Waitlist control receives the adapted 3RP program (3RP-AYA) approximately 2 months after study enrollment.
  Arms: Waitlist Control
Other: 3RP-AYA — The 3RP is a group program that-through a variety of mind-body approaches, such as imagery, relaxation, and yoga-seeks to buffer stress and promote psychological resiliency and physical well-being.
  Arms: 3RP Group Sessions

SUMMARY:
This research study aims to explore the feasibility and acceptability of an adapted resiliency group program, called the Relaxation Response Resiliency Program (3RP-AYA), to reduce stress and promote stress-management among adolescents and young adults who have completed treatment for cancer.

DETAILED DESCRIPTION:
The Relaxation Response Resiliency Program, or 3RP, was developed by researchers at the MGH Benson-Henry Institute for Mind Body Medicine. The 3RP is a group program that-through a variety of mind-body approaches, such as imagery, relaxation, and yoga-seeks to buffer stress and promote psychological resiliency and physical well-being.

The 3RP has not yet been carried out with adolescent or young adult individuals who have recently completed treatment for cancer. As such, the investigators have adapted the original 3RP to target the specific needs of adolescent and young adult patients who are transitioning off active treatment. The investigators are conducting this study to see if the adapted program, the 3RP-AYA, is effective at reducing stress and stress-related symptoms for people of at least age 16 who have completed treatment for cancer within the past five years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with any cancer between ages 14 and 29
* Completed cancer treatment within the past 5 years
* At least 16 years of age at time of enrollment

Exclusion Criteria:

* Unwilling or unable to participate in the study
* Unable to speak or read English
* Is medically or otherwise unable to participate (as determined by a physician or study PI)
* Unwilling or unable to participate in study sessions delivered via the Partners Telehealth videoconferencing software
* Participation in a focus group during Phase 1 (DF/HCC 17-315)

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2025-08-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Giselle K. Perez, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mizrach H, Goshe B, Park ER, Recklitis C, Greer JA, Chang Y, Frederick N, Abrams A, Tower MD, Walsh EA, Huang M, Kenney L, Homans A, Miller K, Denninger J, Usmani GN, Peppercorn J, Perez GK. Randomized Waitlist-Control Trial of a Web-Based Stress-Management and Resiliency Program for Adolescent and Young Adult Cancer Survivors: Protocol for the Bounce Back Study. JMIR Res Protoc. 2022 Jan 26;11(1):e34033. doi: 10.2196/34033. PMID 35080500

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As per our approved protocol, only individuals who signed consent and completed the baseline assessment were considered to be enrolled. Hence, 72 people met this criteria.
Groups:
- 3RP Group Sessions: The 3RP-AYA will be delivered in weekly sessions over the course of approximately 8 weeks, for a total of 8 sessions immediately after enrollment.
- Waitlist Control: The 3RP-AYA will be delivered in weekly sessions over the course of approximately 8 weeks, for a total of 8 sessions 2-months after enrollment.
Period: Overall Study
Arm/Group | 3RP Group Sessions | Waitlist Control
Started (This is total number enrolled (signed consent and completed baseline)) | 35 | 37
Baseline Completion | 35 | 37
Remained Eligible | 33 (n=2 people who were randomized to the intervention had cancer recurrences, causing them to become ineligible.) | 37
Program Initiation | 29 | 35
Follow up Survey #1 | 29 | 35
Follow up Survey #2 | 29 | 34
Completed | 29 | 34
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — Became Ineligible | 2 | 0
Not completed — Missed final survey (3-month follow-up) | 1 | 0
Not completed — Missed final survey (post-treatment | 0 | 1

BASELINE CHARACTERISTICS:
Population: This is a conservative number that consists of all patients who were officially enrolled in the trial (regardless of whether or not they began the intervention), defined as having consented and completed the baseline survey.
Groups:
- Enrolled Patients: All participants who consented and completed the baseline survey
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.76 (3.26)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 18
  Gender: Female | 53
  Gender: Prefer not to describe | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Hispanic or Latino | 15
  Race/ethnicity: Asian | 6
  Race/ethnicity: Black or African American | 3
  Race/ethnicity: White | 43
  Race/ethnicity: Mixed Race | 5
Months since treatment completion [Mean (Standard Deviation); unit: months] | 18.82 (16.06)

OUTCOME MEASURES:

1. Primary Outcome: 3RP-AYA Feasibility: Percent of Identified Eligibles Who Enroll
Description: Percent of identified eligibles who were approached (hence given the opportunity to participate) who enroll (i.e., sign consent and complete baseline). Qualitative information from experts and participants will be used to inform feasibility.
Time Frame: Post-treatment completion (treatment is approximately 8 weeks)
Population: This consists of the total number of individuals who were eligible, were approached and informed about the study, and were offered the opportunity to participate.
Measure: Count of Participants; unit: Participants
Groups:
- Total Individuals Approached: This consists of eligible individuals who were approached and informed about the study (thus had the opportunity to participate)
Arm/Group | Total Individuals Approached
Number analyzed (Participants) | 93
Participants
  Enrolled | 72
  Active refusal | 9
  Passive refusal (made contact but never heard back) | 10
  Interested but unable to make groups | 2

2. Primary Outcome: 3RP-AYA Feasibility: Proportion of Participants Completing the 3RP-AYA Program
Description: Among those who initiated the program, this is the proportion of patients who completed the program (defined as completing 6 out of 8 sessions). Qualitative information from experts and participants will be used to inform feasibility.
Time Frame: Post-treatment completion (treatment is approximately 8 weeks)
Population: Total number of patients who initiated the program.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Completers: Among treatment started, this consists of all participants who completed the 3RP-AYA.
Arm/Group | Treatment Completers
Number analyzed (Participants) | 64
Participants
  Completed 6 out of 8 3RP-AYA sessions. | 55
  Completed less than 6 3RP-AYA | 9

3. Primary Outcome: 3RP-AYA Acceptability: Five Questions
Description: Acceptability will be assessed with five questions rated on a 4-point Likert scale (1=not at all to 4=very). Items will prompt participants to rate the extent to which they found the program to be enjoyable, helpful, applicable, convenient, and satisfaction. Qualitative information from experts and patients will also inform acceptability.
Time Frame: Post-treatment completion (treatment is approximately 8 weeks)
Population: These were inclusive of all responses to the acceptability items.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Completed Post-treatment Survey Acceptability Items: Denominator is the number of individuals who responded to the acceptability measure.
Arm/Group | Completed Post-treatment Survey Acceptability Items
Number analyzed (Participants) | 60
units on a scale
  How enjoyable was the program | 3.62 (.69)
  How helpful was the program? | 3.45 (.75)
  How relevant was the program? | 3.60 (.74)
  How convenient was the program | 3.67 (.71)
  How satisfied are you with the content? | 3.6 (.62)

ADVERSE EVENTS:
Time Frame: Adverse events data was collected from all participants who initiated treatment (n=64) and monitored throughout the duration of the intervention.
Groups:
- Waitlist Control: * The 3RP-AYA will be delivered in weekly sessions over the course of approximately 8 weeks, for a total of 8 sessions
  * Mini relaxation practice
  * Weekly goal check-ins
  * RR-practice
  Waitlist control: The 3RP is a group program that-through a variety of mind-body approaches, such as imagery, relaxation, and yoga-seeks to buffer stress and promote psychological resiliency and physical well-being. Waitlist control receives the adapted 3RP program (3RP-AYA) approximately 2 months after study enrollment.
- 3RP Group Sessions: * The 3RP-AYA will be delivered in weekly sessions over the course of approximately 8 weeks, for a total of 8 sessions
  * Mini relaxation practice
  * Weekly goal check-ins
  * RR-practice
    3RP-AYA: The 3RP is a group program that-through a variety of mind-body approaches, such as imagery, relaxation, and yoga-seeks to buffer stress and promote psychological resiliency and physical well-being.
Arm/Group | Waitlist Control | 3RP Group Sessions
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 0/31 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT03768336/Prot_SAP_000.pdf